CLINICAL TRIAL: NCT06092554
Title: Probiotics in ICU to Reduce Ventilator-Associated Pneumonia: A Double-blind Multicentre Randomized Clinical Trial
Brief Title: Probiotics to Actively Counter Ventilator Associated Pneumonia (PROACT)
Acronym: PROACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Collaborators: Uni-Pharma (Industry)
Responsible Party: Principal Investigator, Filomena Puntillo, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1336/CE-PROACT
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator Associated Pneumonia; Traumatic Brain Injury; stroke; probiotics; VAP; TBI
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Intervention Model Description: The present study will be a multicenter, randomized, double-blind, placebo-controlled trial. Allocation will rely on a computer-based random number generator provided in a sequentially numbered, sealed, opaque envelope.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A numbered sealed envelope will be used to ensure blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional: Probiotics (Experimental): Patients will receive a four probiotic preparation (LactoLevure, UniPharma, Athens, Greece).) in capsules containing: Lactobacillus acidophilus LA-5 [1.75 × 109 colony-forming units (cfu)], Lactobacillus plantarum (0.5 × 109 cfu), Bifidobacterium lactis BB12 (1.75 × 109 cfu) and Saccharomyces boulardii (1.5 × 109 cfu).
  Interventions: Dietary Supplement: LactoLevure
- Control: Placebo (Placebo Comparator): Patients will receive a placebo in capsules containing powdered glucose polymer.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LactoLevure — Patients will receive two capsules, twice daily for 30 days, one through the nasogastric tube and one spread on the oropharynx. The probiotic capsules look identical to the placebo capsules; the powder will be similar when opened. The capsule for nasogastric tube will be opened and suspended in 100 ml of tap water. The capsule for the oropharynx will be opened and suspended in sterile water based surgical lubricant. The administration must happen at least 30 minutes after oral antiseptic product usage (e.g. daily chlorhexidine oral care), which otherwise might neutralize the study supplement's action.
  Arms: Interventional: Probiotics
Other: Placebo — Patients will receive two capsules, twice daily for 30 days, one through the nasogastric tube and one spread on the oropharynx. The placebo capsules contain a powdered glucose polymer that is unharmful for the patient and will be provided by the sponsor. The placebo capsules look identical to the probiotic capsules; the powder will be similar when opened. The capsule for nasogastric tube will be opened and suspended in 100 ml of tap water. The capsule for the oropharynx will be opened and suspended in sterile water based surgical lubricant. The administration must happen at least 30 minutes after oral antiseptic product usage (e.g. daily chlorhexidine oral care), which otherwise might neutralize the study supplement's action.
  Arms: Control: Placebo

SUMMARY:
PROACT study aims to resolve uncertainties to influence actual practice guidelines or public health policing regarding VAP prevention in ICU by using probiotics administration.

Multi-trauma patients with a head injury OR stroke or brain haemorrhage patients without any sign of aspiration and lung infection will be enrolled and randomized to either placebo or probiotic treatment to assess if VAP and mortality can be reduced in the interventional group.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia represents a burden in ICU with a mortality rate approaching 50%. Ventilator-associated pneumonia (VAP) reduction care bundle is a grouping of evidence-based, high-impact interventions.

Among these recommendations:

* raised head of bed (minimizes microaspiration)
* daily sedation hold and assessment of readiness to extubate (decreases length of stay)
* use of subglottic secretion drainage
* avoidance of scheduled ventilator circuit changes
* peptic ulcer prophylaxis (minimizes complications and length of stay)
* venous thrombo-embolism prophylaxis (minimizes complications and length of stay) Probiotics administration does not figure yet in these recommendations despite the literature showing interesting results in VAP reduction, particularly in specific subsets of patients such as trauma. Tsilika et al. demonstrated a VAP reduction in trauma patients with a head injury. The incidence was lowered to 11.9% in the interventional group with a four-probiotic preparation administration from 28.3 % in the placebo group. The same probiotic preparation has been used in multiple trauma patients to reduce surgical site infections, supporting a possibly prophylactic administration of probiotics. A different two-probiotic preparation was given in stroke patients and showed a VAP incidence reduction in the probiotic group. Stroke patients and trauma patients with a head injury share a common pathophysiology, as traumatic brain injury is considered a risk factor for stroke.

Recent reviews and meta-analyses suggest that probiotics administration may reduce VAP incidence, but more studies with a higher level of evidence and low bias are warranted. The rationale for this finding is yet to be understood. Still, it might depend on the communications between the Gut microbiota (GM) and the oral microbiota (OM) on one side and the lung and its microbiota on the other, along the gut-lung and the gut-bone marrow-lung axes. Notably, short-chain fatty acids (SCFAs) such as butyrate, acetate and propionate produced by the GM by fibre fermentation may have anti-inflammatory effects that strengthen the respiratory tract's epithelial barrier. Tailored and early probiotic administration in the critically ill patient when he enters the ICU, may positively modulate the GM and protect the patient from the harmful downside of the GM disruption. The GM imbalance, called dysbiosis, occurs within six hours of ICU admission, leading to lower bacterial diversity and variability while opportunistic pathogens take over symbiotics. Disrupting this vicious cycle which transforms the local GM into a pathobiota, may play a key role in preserving the good functioning of the gut-lung axis. The diversity of the results of published Randomized Controlled Trials (RCT) guiding the necessity for meta-analysis is probably coming from the heterogeneity of the studied patient population and one inclusion bias: it seems that for probiotics to act prophylactically, the enrolled patient population should be as much as possible devoid of any infection. Indeed a recent large-scale RCT from Canada failed to show any benefit of probiotic treatment to reduce the incidence of VAP. However, most participants were already on antibiotics for unspecific infections, and the methods lacked microbiology diagnosis to support VAP detection.

PROACT is a double-blind randomized placebo-controlled clinical trial where the effect of a four probiotic preparation (Lactolevure, Unipharma, Greece) is studied on multi-trauma patients with a head injury OR stroke or brain haemorrhage patients without any sign of aspiration and lung infection to assess whether this supplementation can reduce VAP and mortality.

Patients eligible for enrollment are admitted to the hospital from the emergency department or transferred from another ICU. A legal representative will be asked for written informed consent once a patient classifies as acute brain trauma, stroke, or brain hemorrhage patient. Therefore, eligibility screening can start, and exclusion criteria will first be assessed. If the patient does not meet any exclusion criteria, he will also be considered for inclusion criteria. If the patient meets all the inclusion criteria, he can be successfully enrolled in the study.

The patient will be blindly assigned at a 1:1 ratio to either the interventional (probiotics) group or the control ( placebo) group.

The research coordinator and the sub-investigators will assess patients daily in the ICU, where most data will be gathered. The investigators and the clinicians evaluating the patients will be blind to the allocated treatment for the entire study duration.

This includes:

1. Baseline data: demographics (age, gender, height, weight, country of origin), total comorbidities number on admission, cardiovascular axis on admission, pulmonary axis on admission, metabolic axis on admission, liver axis on admission, rheumatic axis on admission, renal axis on admission, neurologic axis on admission, history of smoking, Glasgow Coma Scale (GCS) on admission, sequential organ failure assessment (SOFA) score on admission, Acute Physiology and Chronic Health Evaluation (APACHE II) score on admission, Simplified Acute Physiology Score (SAPS) II score on admission, Charlson Comorbidity Index. Before start of the study drug, one sample of tracheobronchial secretions will be collected and analyzed quantitatively. This step is necessary to define the modified intention-to-treat (mITT) population.
2. Daily data: vital signs, sepsis, septic shock, CRBSI, Catecholamine support, Enteral feeding, Parenteral feeding, Enteral + Parenteral feeding, prokinetics, beta-lactamase inhibitor, second-generation cephalosporin, third-generation cephalosporin, piperacillin/tazobactam, metronidazole, clindamycin, amikacin, glycopeptide, microbiology and antibiogram (if available), GCS score, SOFA score, diarrhoea (type 6/7 bristol stool chart), mechanical ventilation, Oxygen saturation (SpO2), culture results, adverse events.
3. VAP screening: every day, the patient will be screened explicitly for VAP by the attending physician. The screening protocol begins with clinical suspicion. The presence of new or progressive radiographic infiltrates and at least two of three clinical criteria [19] ( fever/hypothermia, leukocytosis/leukopenia, purulent secretions) represent the protocol trigger. Leukocytosis is defined as an elevation in the absolute White Blood Cells (WBC) count (10,000 cells/μL), while leukopenia is defined as a reduction in the WBC count (<3500 cells/μL) [20]. Hypothermia is defined as a body core temperature of <35.0 °C (95.0 °F) [21], while fever is defined as a body core temperature of ≥38.3°C (101° F) [22]. Once the clinical suspicion is realized, samples of respiratory secretions, i.e. tracheal aspirate and bronchoalveolar lavage (BAL), are obtained non-invasively. Samples will be quantitatively cultured at the local hospital laboratory. Part of the samples will be stored at -20 °C and shipped by air transport to the Laboratory of Immunology of Infectious Diseases of the 4th Department of Internal Medicine of ATTIKON University General Hospital (124 62 Athens, Greece) for molecular testing. A VAP diagnosis will be established if either quantitative cultures yield more than 105 cfu/ml growth of one pathogen or when more than 104 copies of a pathogen are grown in molecular testing.

FOLLOW-UP: The data collection will continue for at least 30 days unless the patient is successfully extubated, interrupting mechanical ventilation. In this case, the data collection and the probiotic administration will continue for 72 hours after successful weaning to pass the time window for a late VAP diagnosis. The data collection will continue for two additional days if a patient is still in the ICU after the thirtieth day until discharge, although the intervention stops. If VAP is diagnosed, the patient will continue the probiotic administration for up to 30 days as per the study protocol since there may still be a beneficial effect on the secondary outcomes.

Biological samples will be collected pre- and post-treatment (after 30 days or 72h after successful extubation) to study how probiotics administration affects GM's composition. The samples are going to be faeces, blood and urine.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-80 years
* at least one of the following conditions: a) recent trauma involving head injury and at least one more organ system; b) stroke or brain hemorrhage without any sign of aspiration and lung infection
* intubation and start of mechanical ventilation. This needs to start immediately after the event described in the inclusion criteria (b). For cases of head trauma this is defined as start in the ambulance or the emergency department
* likelihood that the duration of mechanical ventilation would be at least six days
* written informed consent provided by the patient or legal representative

Exclusion Criteria:

* has received mechanical ventilation more than 72 hours from start of screening
* pregnancy or Lactation
* patients at risk of iatrogenic probiotic infection e.g. immunosuppression which includes
* HIV <200 CD4 cells/μL
* those receiving chronic immunosuppressive medications (e.g., azathioprine, cyclosporine, cyclophosphamide, tacrolimus, methotrexate, mycofenolate, Anti-IL2)
* previous transplantation at any time
* malignancy requiring chemotherapy in the last 3 months
* neutropenia [absolute neutrophil count < 500])
* patients with a primary diagnosis of severe pancreatitis (Ranson score of 3 or more). Mild and moderate pancreatis is not excluded
* ischemic bowel disease
* oropharyngeal mucosal injury
* inability to receive enteral medications
* intent to withdraw advanced life support as per ICU doctor in charge
* patients at risk of endovascular infection which includes

  1. previously documented rheumatic heart disease, congenital valve disease, surgically repaired congenital heart disease, unrepaired cyanotic congenital heart disease, any intracardiac repair with prosthetic material [mechanical or bioprosthetic cardiac valves]
  2. previous or current endocarditis
  3. permanent endovascular devices (e.g., endovascular grafts [e.g., aortic aneurysm repair, stents involving large arteries such as aorta, femorals and carotids] inferior vena cava filters, dialysis vascular grafts
  4. tunnelled (not short-term) hemodialysis catheters
  5. pacemakers or defibrillators

     Patients with peripherally inserted central catheters (PICCs), temporary central venous catheters, central venous dialysis catheters, coronary artery stents, coronary artery bypass grafts (CABG), or neurovascular coils are not excluded, nor are patients with mitral valve prolapse or bicuspid aortic valve if they do not meet any other exclusion criteria.
* patients with sepsis and/or septic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Vap Incidence | 45 days
  VAP is defined as first episode of lower respiratory tract infection that meets all the following criteria: (a) onset >48 h after initiation of mechanical ventilation; (b) increase in SOFA score by ≥1 point; (c) new infiltrate in chest X-ray or chest computed tomography; (d) core temperature >38°C; (e) purulent tracheobronchial secretions; (f) clinical pulmonary infection score (CPIS) >6 ; and (g) isolation of a pathogen from BAL fluid (>1 × 104 cfu/mL) or tracheal aspirate (>1 × 105 cfu/mL) . This is analyzed for the ITT population. The ITT comprises the total of enrolled and randomized patients.

SECONDARY OUTCOMES:
Vap incidence analyzed for mITT | 45 days
  The mITT comprised only patients with less than 102 cfu/ml of bacterial growth in tracheobronchial secretions before start of the study drug.
Sepsis | 45 days
  Sepsis is defined as a new infection with at least a 2-point increase in the total SOFA score.
  The endpoint will be analyzed for both the ITT and mITT populations.
Septic shock | 45 days
  Septic shock is defined as sepsis aggravated by hypotension and serum lactate level >2 mmol/L (18 mg/dL) that requires vasopressors administration despite adequate volume resuscitation.
  The endpoint will be analyzed for both the ITT and mITT populations.
Catheter-related bloodstream infections (CRBSI) | 45 days
  CRBSI, according to the Infectious Diseases Society of America, is defined when one of the following criteria is met 1) Isolation of the same pathogen from a quantitative blood culture drawn through the central line and from a peripheral vein with the single bacterial colony count at least threefold higher in the sample from the central line as compared to that obtained from a peripheral vein 2) same organism recovered from percutaneous blood culture and from quantitative (>15 colony-forming units) culture of the catheter tip 3) a shorter time to positive culture (>2 hours earlier) in the central line sample than the peripheral sample (differential time to positivity [ DTP ]).
  The endpoint will be analyzed for both the ITT and mITT populations.
ICU length of stay | 45 days
  Duration in days of the patient stay in the ICU. The endpoint will be analyzed for both the ITT and mITT populations.
Mechanical ventilation days | 45 days
  Mechanical ventilation days is to be intended as the total number of days during which the patient underwent mechanical ventilation.
  The endpoint will be analyzed for both the ITT and mITT populations.

CONTACTS AND LOCATIONS:
Overall Officials: Filomena Puntillo, MD, PhD, Study Director — University of Bari; Alberto Corriero, MD, Principal Investigator — University of Bari
Locations (9):
- Hospital Erasme, Brussels, Belgium
- Italy (8):
  - Regional General Hospital F. Miulli, Acquaviva delle Fonti, BA
  - Intensive Care Unit, Policlinico di Bari, Bari, BA
  - Azienda Ospedaliero Universitaria di Alessandria SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Di Venere, Bari
  - AUSL Bologna Ospedale Bellaria, Parma
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda ospedaliera Santa Maria di Terni, Terni

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corriero A, Soloperto R, Giglio M, Salvagno M, Trerotoli P, Grasso S, Ribezzi M, Mosca A, Petrillo C, De Toma N, Magnesa G, Giacomucci A, Accattoli R, Gadaleta RM, Florio M, Cariello M, Moschetta A, Puntillo F, Taccone FS, Ranieri VM. Probiotics to reduce ventilator-associated pneumonia in adults with acute non-anoxic brain injury: Study Protocol for a Double-Blind Multicenter Randomized International Clinical Trial (PROACT). Trials. 2025 Nov 10;26(1):484. doi: 10.1186/s13063-025-09230-w. PMID 41214813